CLINICAL TRIAL: NCT02261415
Title: The HeLiX (Hemorrhage During Liver Resection: traneXamic Acid) Trial: Tranexamic Acid (TXA) Versus Placebo to Reduce Perioperative Blood Transfusion in Patients Undergoing Liver Resection: A Randomized Controlled Trial
Brief Title: The HeLiX (Hemorrhage During Liver Resection: traneXamic Acid) Trial
Acronym: HeLiX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: HepatoPancreaticoBiliary (HPB) Concept Team (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 244-2014
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cancer; Tumour; Surgery
Keywords: blood transfusion; blood loss; feasibility; outcome; liver resection
MeSH Terms: conditions — Neoplasms; Hemorrhage | interventions — Tranexamic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (TXA) (Experimental): 1 g TXA bolus injection + 1 g TXA infusion from induction over 8 hours
  Interventions: Drug: Tranexamic acid (TXA)
- Normal saline (0.9% sodium chloride) (Placebo Comparator): 1 g saline bolus injection + 1 g saline infusion from induction over 8 hours
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — 1 g TXA bolus injection + 1 g TXA infusion from induction over 8 hours
  Other Names: Cyklokapron
  Arms: Tranexamic acid (TXA)
Drug: Normal saline — 1 g saline bolus injection + 1 g saline infusion from induction over 8 hours
  Other Names: 0.9% sodium chloride
  Arms: Normal saline (0.9% sodium chloride)

SUMMARY:
This is a Phase III multicentre randomized controlled trial (RCT) to evaluate the impact of tranexamic acid (TXA) on perioperative blood transfusion in patients undergoing liver resection. The rationale for this study includes: (1) experimental evidence supporting the use of TXA in other surgical populations; (2) lack of evidence in patients undergoing liver resection; (3) clinical uncertainty and extensive support amongst hepatobiliary surgeons, anaesthesiologists, and hematologists for this proposed trial; (4) a feasible and efficient study design; and (5) the importance of the question: incidence of blood transfusion in patients undergoing liver resection is high, and the consequences serious. The sample size for this study is 1230 participants.Participants enrolled in the prior Vanguard study will proceed directly into the RCT.

DETAILED DESCRIPTION:
Purpose Compelling biological rationale and indirect evidence from other settings suggest that there is potential benefit to administering TXA to patients undergoing liver resection. A lack of consensus in the hepatobiliary community and lack of direct evidence in patients undergoing liver resection mandate a RCT.

Hypothesis To determine the impact of perioperative administration of TXA to patients undergoing liver resection on the need for blood transfusion and long-term survival.

Justification If TXA use in liver resection resulted in an important decrease in blood transfusions, clinical practice worldwide would be likely to change. Over 2000 patients in Canada undergo liver resection annually and could benefit from this simple, low-cost intervention. This intervention could easily be implemented in other countries, where many more patients undergo liver resection annually. Furthermore, TXA may be beneficial in other operative fields where bleeding is a major problem, including thoracic surgery, colorectal surgery, and many others.

Objectives

The primary outcome of the RCT will be:

1) Receipt of blood transfusion (% transfused): 7 days

The secondary outcomes of the RCT are:

1. Intraoperative blood loss will be assessed by adding the net weight of sponges and fluid suction (minus irrigation and intraoperative bile or other fluids in suction/sponge)
2. Total blood loss (postoperative day (POD)0 - POD7) will be assessed by Gross' formula, which uses the maximum postoperative decrease in the level of hemoglobin adjusted for the weight and height of the patient
3. Number of packed red blood cells (PRBC) units transfused (POD0 - POD7)
4. Postoperative incidence of symptomatic venous thromboembolic event confirmed with either computed tomography (CT) angiogram (for pulmonary embolism) or venous Doppler ultrasound (for deep venous thrombosis) (within 90 days of surgery)
5. Postoperative complications (within 90 days of surgery) will be determined using the Clavien-Dindo classification
6. Recurrence free survival (within 5 years of surgery) will be determined by review of patient medical record every 6 months until 5 years post-surgery

   a. Recurrence free survival is defined as the time from POD0 to the first event that is recurrent (local or distal) cancer or death (from any cause)
7. Overall survival (within 5 years of surgery) will be determined by review of patient medical record every 6 months until 5 years post-surgery

   a. Overall survival is defined as the time from date of POD0 to death from any cause
8. QOL will be determined by administering European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) -C30 and the QLQ- Liver Metastases Colorectal (LMC) 21 at baseline, 30 and 90 days following surgery
9. Perioperative mortality will be recorded between POD0 and POD7
10. Economic analysis will assess impact of TXA incorporation on health care resources and strategies for systematic utilization of TXA

Research Method This is a Phase III multicentre randomized controlled trial (RCT) to evaluate the impact of tranexamic acid (TXA) on perioperative blood transfusion in patients undergoing liver resection. The trial will conceal allocation, maximize possible blinding, independently assess the appropriateness of transfusion, use strategies to limit loss to follow-up and crossovers, and use a conservative stopping rule. Patients will be administered a single dose of study drug intravenously immediately after induction of anaesthesia, followed by infusion over eight hours.

Statistical Analysis Primary analysis will include only patients who underwent liver resection; patients who are randomized but do not receive liver resection (usually due to more advanced disease identified intraoperatively) will be excluded. A sensitivity analysis will be conducted whereby all randomized patients are included in the assessment of the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open or laparoscopic liver surgery
* Age ≥18 years
* Cancer related diagnosis or indication (e.g. pre-cancer, suspicion of cancer, definite cancer)

Exclusion Criteria:

* Severe anemia (hemoglobin (Hgb) levels <90 g/l)
* Documented arterial or venous thrombosis at screening or in past three months (not including therapeutic portal vein embolization)
* Anticoagulants (other than low-molecular-weight heparin (LMWH) or heparin in prophylactic doses to prevent deep vein thrombosis), direct thrombin inhibitors or thrombolytic therapy administered or completed within last week
* Known disseminated intravascular coagulation
* Severe renal insufficiency (creatinine clearance (CrCl) <30 ml/min)
* History of seizure disorder
* Pregnant or lactating (a negative urine pregnancy test must be obtained for women of child bearing potential during the pretreatment evaluation)
* Acquired disturbance of colour vision
* Hypersensitivity to TXA or any of the ingredients
* Unable to receive blood products (i.e. difficulty with cross matching, refuses blood transfusion, or a past history of unexplained severe transfusion reaction)
* Previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1386 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Receipt of blood transfusion (% transfused): 7 days | 7 days
  Receipt of one or more RBC transfusions between Day 0 and Day 7

SECONDARY OUTCOMES:
Intraoperative blood loss | 7 days
  Intraoperative blood loss will be assessed by adding the net weight of sponges and fluid suction (minus irrigation and intraoperative bile or other fluids in suction/sponge)
Total blood loss | 7 days
  Total blood loss (postoperative day (POD)0 - POD7) will be assessed by Gross' formula, which uses the maximum postoperative decrease in the level of hemoglobin adjusted for the weight and height of the patient
Number of packed red blood cells (PRBC) units transfused | 7 days
  Number of packed red blood cells (PRBC) units transfused (POD0 - POD7)
Postoperative incidence of symptomatic venous thromboembolic event | 90 days
  Postoperative incidence of symptomatic venous thromboembolic event confirmed with either computed tomography (CT) angiogram (for pulmonary embolism) or venous Doppler ultrasound (for deep venous thrombosis) (within 90 days of surgery)
Postoperative complications assessed using Clavien-Dindo Grading System | 90 days
  Postoperative complications (within 90 days of surgery) will be determined using the Clavien-Dindo classification
Recurrence Free Survival (within 5 years of surgery) | 60 months
  Disease recurrence is defined as the clinical presence of cancer that has either been confirmed by biopsy, has had treatment initiated, or is documented in the treating physician's notes. Five year disease recurrence from day of surgery will be evaluated approximately every 6 months until 5 years via medical record review.
Overall Survival (within 5 years of surgery) | 60 months
  Overall survival is defined as the time from date of surgery to death from any cause. It will be determined by review of patient medical record every 6 months until 5 years post-surgery.
Quality of Life (QOL) Assessment using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | Baseline, 30 days, 90 days
  QOL will be determined by administering the EORTC QLQ-C30 at baseline, 30 and 90 days following surgery.
Quality of Life (QOL) Assessment using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Liver Module (LM)C21 Questionnaire | Baseline, 30 days, 90 days
  QOL will be determined by administering QLQ-LMC21 at baseline, 30 and 90 days following surgery.
Perioperative mortality | 7 days
  Perioperative mortality will be recorded between POD0 and POD7
Compare the cost of tranexamic acid (TXA) versus placebo on perioperative blood transfusion in patients undergoing liver resection | 90 days
  Economic analysis will assess impact of TXA incorporation on health care resources and strategies for systematic utilization of TXA. The analysis will be using data collected in the randomized controlled trial from a societal perspective.The output of the economic analysis is the incremental cost of TXA compared to placebo (control group).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (11):
- Mayo Clinic, Rochester, Minnesota, United States
- Canada (10):
  - Foothills Hospital, Calgary, Alberta
  - Kelowna General Hospital, Kelowna, British Colombia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Health Research Institute, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karanicolas PJ, Lin Y, McCluskey SA, Tarshis J, Thorpe KE, Wei A, Dixon E, Porter G, Chaudhury P, Nanji S, Ruo L, Tsang ME, Skaro A, Eeson G, Cleary S, Moulton CA, Ball CG, Hallet J, Coburn N, Serrano PE, Jayaraman S, Law C, Tandan V, Sapisochin G, Nagorney D, Quan D, Smoot R, Gallinger S, Metrakos P, Reichman TW, Jalink D, Bennett S, Sutherland F, Solano E, Molinari M, Tang ES, Warner SG, Bathe OF, Barkun J, Kendrick ML, Truty M, Roke R, Xu G, Lafreniere-Roula M, Guyatt G; HPB CONCEPT Team. Tranexamic Acid in Patients Undergoing Liver Resection: The HeLiX Randomized Clinical Trial. JAMA. 2024 Oct 1;332(13):1080-1089. doi: 10.1001/jama.2024.11783. PMID 39158894
- [Derived] Karanicolas PJ, Lin Y, McCluskey S, Roke R, Tarshis J, Thorpe KE, Ball CG, Chaudhury P, Cleary SP, Dixon E, Eeson G, Moulton CA, Nanji S, Porter G, Ruo L, Skaro AI, Tsang M, Wei AC, Guyatt G; HepatoPancreaticoBiliary Community of Surgical ONcologists: Clinical, Evaluative, and Prospective Trials (HPB CONCEPT) Team. Tranexamic acid versus placebo to reduce perioperative blood transfusion in patients undergoing liver resection: protocol for the haemorrhage during liver resection tranexamic acid (HeLiX) randomised controlled trial. BMJ Open. 2022 Feb 24;12(2):e058850. doi: 10.1136/bmjopen-2021-058850. PMID 35210348